CLINICAL TRIAL: NCT03567954
Title: The Diagnostic Accuracy of Ultrasound in Detecting Rotator Cuff Tears in Patients Who Sustained a Proximal Humerus Fracture
Brief Title: The Accuracy of Ultrasound in Detecting Rotator Cuff Tears in Proximal Humerus Fracture Patients
Status: Terminated | Type: Observational
Why Stopped: Low inclusionrate due to logistic challenges
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Viborg, Skive (Other); Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ProxHumUS
Record Dates: First submitted 2018-05-25; First posted 2018-06-26 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2022-12

CONDITIONS: Rotator Cuff Tear; Proximal Humeral Fracture
Keywords: Diagnostic ultrasound
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound examination of the rotator cuff tendons — An ultrasound scan of the rotator cuff tendons will be performed to determine the presence of a rotator cuff tear or not

SUMMARY:
The aim of this study is to determine the diagnostic accuracy of ultrasonography (US) in detecting full-thickness (a lesion that extends through both the bursal and articular part of the tendon) rotator cuff tear in patients who have sustained a proximal humerus fracture, using operative examination as the golden standard.

DETAILED DESCRIPTION:
Although most of the focus concerning proximal humerus fractures is on the bony structures, injuries in the musculotendinous insertion regions of the rotator cuff musculature may also need attention in the treatment. Ultrasound is a painless and non-invasive screening modality in patients with a suspected rotator cuff tear. It is a user-dependent modality and health professionals must possess the competence and training before using it. To the investigators knowledge, no studies have investigated the accuracy of ultrasound in detecting rotator cuff tears, in patients who sustained a proximal humerus fracture.

ELIGIBILITY:
Inclusion Criteria:

* Displaced proximal humeral fracture
* Referred to operative treatment

Exclusion Criteria:

* Younger than 18 years old
* Non-independent
* Does no understand written and spoken guidance in local language, Danish, Swedish or Finnish
* Open fracture
* Isolated tuberculum fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults referred to Viborg Regional Hospital and Tampere University Hospital, Finland, under suspicion of a proximal humerus fracture.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Full-thickness rotator cuff tear in the shoulder | Ultrasound scan is performed once; Baseline (prior to operation which is the golden standard)
  The outcome is dichotomous; yes/no and will be used to estimate the sensitivity, specificity, the negative predictive value and the positive predictive value

SECONDARY OUTCOMES:
Partial-thickness rotator cuff tear in the shoulder | Ultrasound scan is performed once; Baseline (prior to operation which is the golden standard)
  The outcome is dichotomous; yes/no and will be used to estimate the sensitivity, specificity, the negative predictive value and the positive predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Helle Østergaard, MSc., PhD student, Principal Investigator — Viborg Regional Hospital
Locations (2):
- Viborg Regional Hospital, Viborg, Denmark
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No